CLINICAL TRIAL: NCT01957709
Title: A Pilot Study to Test Whether Systemic Interferon Gamma Increases Tumor Class I MHC Expression in Patients With Synovial Sarcoma and Myxoid/Round Cell Liposarcoma
Brief Title: Recombinant Interferon Gamma in Treating Patients With Soft Tissue Sarcoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enough samples were collected for data analysis.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Horizon Pharma USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2705.00; NCI-2013-01779 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2705 (Other: Fred Hutchinson Cancer Research Center); 2705.00 (Other: Fred Hutch/University of Washington Cancer Consortium); K12CA076930 (NIH); K23CA175167 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Myxoid Liposarcoma; Round Cell Liposarcoma; Synovial Sarcoma
MeSH Terms: conditions — Liposarcoma, Myxoid; Sarcoma, Synovial | interventions — Interferon-gamma

STUDY DESIGN:
Intervention Model Description: 100 mcg/m2 weekly injection for four weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Basic science (interferon gamma and MHC expression) (Experimental): Patients receive recombinant interferon gamma subcutaneously weekly for 4 weeks before surgery.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Recombinant Interferon Gamma

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Recombinant Interferon Gamma — Given subcutaneously weekly for four weeks prior to surgery.
  Other Names: Gamma Interferon (GEN); Gamma Interferon-SCH; Gamma-Interferon; Ginterferon; IFN-g; Interferon Gamma; Interferon Gamma (BIO); Interferon, Gamma

SUMMARY:
This pilot clinical trial studies the effect of recombinant interferon gamma on tissue in treating patients with soft tissue sarcoma. Interferon gamma may interfere with the growth of tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether systemic administration of interferon (IFN) gamma (recombinant interferon gamma) will increase class I major histocompatibility complex (MHC) expression in synovial sarcoma (SS) and myxoid/round cell liposarcoma (MRCL) tumors.

SECONDARY OBJECTIVES:

I. To determine whether systemic administration of IFN gamma will increase class II MHC expression in SS and MRCL tumors.

II. To examine changes in the immune response to MRCL and SS by examining changes in the immune infiltrates, antibody response and antigen specific T cell response before and after IFN gamma treatment.

OUTLINE:

Patients receive recombinant interferon gamma subcutaneously (SC) every 7 days for 4 weeks before surgery.

After completion of study, patients are followed up at 2 weeks post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of synovial sarcoma and myxoid/round cell liposarcoma
2. Male or female subject, 18 or older
3. A superficial tumor easily and safely accessible for a research biopsy or are being considered for resection or biopsy of their tumor as part of standard of care and have recent pathology.
4. Zubrod performance status of '0-2' or Karnofsky score > 60%
5. No treatment with systemic anti-cancer treatment (chemotherapy or biologics) within 2 weeks of starting interferon gamma
6. Patients with a history of coronary artery disease must have had a normal stress test within 180 days of starting IFN gamma
7. Must have been off metformin for at least 2 weeks prior to starting IFN gamma
8. No use of full dose, therapeutic anti-coagulation. However, low dose warfarin for catheter prophylaxis or acetylsalicylic acid are acceptable.
9. No thrombotic event within 6 months (deep vein thrombosis, pulmonary embolism) of starting IFN gamma

Exclusion Criteria:

1. Active infection requiring oral or intravenous antibiotics
2. Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception or abstinence. Women of childbearing potential must have a negative pregnancy test within two weeks prior to entry.
3. Serum creatinine > 1.5 mg/dL or Glomerular Filtration Rate < 50
4. Significant hepatic dysfunction (SGOT > 150 IU or > 3x upper limit of normal; bilirubin > 1.6 mg/dL; prothrombin time > 1.5x control).
5. Known central nervous system (CNS) metastasis. Once CNS metastasis have been treated these patients may participate if they are otherwise good trial candidates.
6. Current treatment with steroids (must be discontinued 1 week before starting IFN gamma)
7. Hemoglobin A1C > 8.5%
8. Uncontrolled hypertension, blood pressure (BP) > 150/100 mmHg; patients with elevated BP may enroll once BP is corrected
9. Cancer/testis antigen 1B (NY-ESO-1) specific T cell therapy within 1 year of starting on the trial
10. New (< 6 months) cardiac arrhythmia (electrocardiogram [EKG] should be performed within 2 weeks of starting IFN gamma).
11. History of clinically significant congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Pollack, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroeder BA, Black RG, Spadinger S, Zhang S, Kohli K, Cao J, Mantilla JG, Conrad EU, Riddell SR, Jones RL, Yee C, Pollack SM. Histiocyte predominant myocarditis resulting from the addition of interferon gamma to cyclophosphamide-based lymphodepletion for adoptive cellular therapy. J Immunother Cancer. 2020 Apr;8(1):e000247. doi: 10.1136/jitc-2019-000247. PMID 32269142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done in the Seattle Cancer Care Alliance medical clinic, or by patient referral.
Groups:
- Basic Science (Interferon Gamma and MHC Expression): Patients receive recombinant interferon gamma SC weekly for 4 weeks before surgery.
  Laboratory Biomarker Analysis: Correlative studies
  Recombinant Interferon Gamma: Given Subcutaneously
Period: Overall Study
Arm/Group | Basic Science (Interferon Gamma and MHC Expression)
Started | 8
Completed | 7
Not Completed | 1
Not completed — Patient refused to complete post-tx bx | 1

BASELINE CHARACTERISTICS:
Groups:
- Basic Science (Interferon Gamma and MHC Expression): Patients receive recombinant interferon gamma SC every 7 days for 4 weeks before surgery or thrice weekly for 2 weeks before surgery.
  Laboratory Biomarker Analysis: Correlative studies
  Recombinant Interferon Gamma: Given SC
Arm/Group | Basic Science (Interferon Gamma and MHC Expression)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Class I Major Histocompatibility Complex (MHC) Expression After Treatment With IFN Gamma
Description: It would be highly relevant to observe marked increase macrophages (effect size > 2.5). Four patients gives over 90% power to detect such a large increase with a two-tailed alpha of 0.05.
Time Frame: Baseline to up to 2 weeks post-surgery
Measure: Median (Full Range); unit: percentage of MHC Class I+ on tumor cell
Arm/Group | Basic Science (Interferon Gamma and MHC Expression)
Number analyzed (Participants) | 8
percentage of MHC Class I+ on tumor cell
  Pre-treatment | 8.91 [.131 to 51.6]
  Post-treatment | 26.6 [1.39 to 92.2]

2. Secondary Outcome: MHC Class II Expression
Description: To determine whether systemic administration of IFNg will increase class II MHC expression in SS and MRCL tumors.
Time Frame: Baseline to 2 weeks post biopsy.
Measure: Median (Full Range); unit: percentage of MHC Class II on tumor cell
Arm/Group | Basic Science (Interferon Gamma and MHC Expression)
Number analyzed (Participants) | 8
percentage of MHC Class II on tumor cell
  Pre-treatment | 2.556 [0.0 to 6.10]
  Post-treatment | 6.125 [0.0 to 10.5]

3. Secondary Outcome: Changes in Immune Response
Description: To examine changes in the immune response to MRCL and SS by examining changes in the immune infiltrates, antibody response and antigen specific T cell response before and after IFNg treatment.
Time Frame: Baseline to 2 weeks post biopsy
Measure: Median (Full Range); unit: percentage of T cells
Arm/Group | Basic Science (Interferon Gamma and MHC Expression)
Number analyzed (Participants) | 8
percentage of T cells
  Pre-treatment | 0.14 [0.015 to 1.05]
  Post-treatment | 0.82 [0.074 to 3.39]

ADVERSE EVENTS:
Time Frame: Patients will be evaluated at their baseline visit prior to administration of the IFNg through two weeks following their surgery. Ideally this will be a period of 6-10 weeks, depending on the number of times a patient received IFNg subcutaneously and when their surgery was scheduled.
Arm/Group | Basic Science (Interferon Gamma and MHC Expression)
All-Cause Mortality (participants affected / at risk) | 7/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basic Science (Interferon Gamma and MHC Expression) (N=8)
Flu-like symptoms (General disorders) | 5 (5) — Grade 1: all events
Fatigue (General disorders) | 5 (5) — Grade 1: 4 events Grade 2: 1 event
Chills (General disorders) | 4 (4) — Grade 1: all events
Headache (Nervous system disorders) | 4 (4) — Grade 1: all events
Fever (General disorders) | 2 (2) — Grade 1: all events
Body Aches (Musculoskeletal and connective tissue disorders) | 2 (2) — Grade 1: all events
Injection site pain (General disorders) | 2 (2) — Grade 1: all events
Dizziness (Nervous system disorders) | 1 (1) — Grade 1
Insomnia (Psychiatric disorders) | 1 (1) — Grade 1
Night Sweats (General disorders) | 1 (1) — Grade 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1
Malaise (General disorders) | 1 (1) — Grade 1
Paresthesia (Nervous system disorders) | 1 (1) — Grade 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1
Injection site erythema (General disorders) | 1 (1) — Grade 1
Dry mouth (Gastrointestinal disorders) | 1 (1) — Grade 1
Upper Respiratory Infection (Infections and infestations) | 1 (1) — Grade 2
Diarrhea (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) — Grade 3
Biopsy site pain (General disorders) | 1 (1) — Grade 2

LIMITATIONS AND CAVEATS:
Early termination of trial due to collection of enough data necessary to complete analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT01957709/Prot_SAP_000.pdf